CLINICAL TRIAL: NCT04215237
Title: A Clinical Observational Trail on Atorvastatin Regulates Intestinal Flora and Metabolomics.
Brief Title: How Atorvastatin Affects the Gut Flora and Metabolomics?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: XJTU1AF2018LSK-91
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis | interventions — Atorvastatin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atorvastatin regulates intestinal flora (Other)
  Interventions: Drug: Atorvastatin 20 Mg Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin 20 Mg Oral Tablet — Atorvastatin 20mg oral once a day

SUMMARY:
Recent studies suggest that gut microbiome, the microbial community in the intestine, may directly and indirectly influence the progression of atherosclerosis. The imbalance of gut microbiome may directly promote the formation of atherosclerotic plaques by promoting the inflammatory reaction and oxidative stress affecting vascular endothelial function and increasing platelet activity. Meanwhile, it can indirectly increase the risk of atherosclerosis by enhance insulin resistance, reducing the production of bile acids and raising serum LDL-C and angiotensin levels. As shown in these researches, gut microbiome, acting as a bridge between metabolism, energy and inflammatory responses, may play an important role in cardiovascular diseases, and we believe that the interaction between microbiome and host should be considered in the ASCVD study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years;
* Statin indications such as lipid metabolism disorders, diabetes, elevated CRP, atherosclerosis; stratification according to ASCVD risk; indications for statin treatment
* Not using statins and other lipid-lowering drugs for at least 6 months before enrollment;
* Agree to receive research treatment plan;
* Voluntarily sign the informed consent.

Exclusion Criteria:

* People with active gastrointestinal bleeding or have a clear history of gastrointestinal ulcers or bleeding in the past 2 years;
* Severe renal insufficiency (eGFR <30ml / min / 1.73m2);
* Active hepatitis, liver cirrhosis, or ALT increase more than 3 times;
* Those with severe hypertension (> 180 / 110mmHg) and currently have no control;
* Hemoglobin <100g / L;
* Platelet count <100 × 109 cells / L;
* Suffering from a known serious progressive disease (such as a malignant tumor) or a disease that causes the patient to fail extremely, the estimated survival time is <12 months;
* pregnant or intending to become pregnant;
* Any situation that may interfere with the research process, such as dementia, paralysis, alcoholism, etc .;
* Expected to undergo surgery within 1 year;
* Patients participating in other ongoing clinical studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-13 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of flora | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Zuyi Yuan, Professor, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No